CLINICAL TRIAL: NCT00592436
Title: A Screening Protocol for Children and Adolescents With Attention Deficit Hyperactivity Disorder
Brief Title: Screening Protocol for Children and Adolescents With Attention Deficit Hyperactivity Disorder
Status: Terminated | Type: Observational
Why Stopped: New protocol developed for recruitment of children for all child studies
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Chief, Clinical and Research Programs in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Other Study IDs: 2003-P-000239
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Pediatric ADHD
Keywords: ADHD; pediatric; children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The objective of this protocol is to establish a comprehensive screening process to evaluate the eligibility of potential pediatric subjects for appropriate ADHD clinical research studies.

DETAILED DESCRIPTION:
The ADHD Clinical Research Program at Massachusetts General Hospital currently offers a range of protocols addressing different aspects of ADHD in children and adolescents. Although these protocols have received prior IRB approval, potential participants present with a widely varied set of complaints not always discernable in a telephone screening interview. This state of affairs often makes it difficult to ask subjects and their parents to sign a specific protocol's consent form without obtaining additional clinical information. Because of this, we are proposing that potential subjects and their parents undergo an in-depth clinical assessment that will allow them to be screened by a clinician for eligibility to a diverse clinical research program.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages 6-17
2. Family/guardian contacting the Clinical Research Program in Pediatric Psychopharmacology, with concerns regarding ADHD symptoms in his/her child

Exclusion Criteria:

1. History of significant head trauma with loss of consciousness, organic brain disorders, seizures, or neurological intervention
2. Any significant medical condition, in the judgment of the investigator
3. Mental retardation
4. Pregnancy or lactation
5. Subjects with current, uncontrolled (within the past 3 months) illicit drug or alcohol dependence
6. Sensory difficulties such as deafness or blindness

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with symptoms of ADHD
Sampling Method: Non-Probability Sample
Enrollment: 663 (Actual)
Dates: Start 2003-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Screening Protocol | Screening
  This is a prescreening for potential participation in research studies.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://massgeneral.org/pediatricpsych/home.html